CLINICAL TRIAL: NCT03652311
Title: Pilot Investigation of at Home Caloric Vestibular Neuromodulation for Use in Substance Use Disorders
Brief Title: Investigating the Efficacy of Caloric Vestibular Stimulation in the Treatment of Substance Use Disorders
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Suspended temporarily due to staff changes
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00052544
Record Dates: First submitted 2018-08-17; First posted 2018-08-29 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-08

CONDITIONS: Substance Use Disorders
Keywords: opiate use disorder; neuromodulation; caloric vestibular stimulation; adjunct therapy
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: This study is designed as a nonrandomized, single-blind, sham-controlled trail in which willing participants will receive a 5 day course of twice daily caloric vestibular stimulation (CVS) or sham treatment
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know if they are receiving therapeutic CVS or sham stimulation.
  Participant survey responses will be blinded during analysis and only the use of non-informative catalogue will be used. This will eliminate bias in the analysis of the survey data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TNM Device Group (Experimental): In this arm participants will receive 5 sessions of twice daily treatments of 15 minutes of caloric vestibular stimulation (CVS) using the ThermoNeuroModulation TNM Device. In addition, participants will continue with the standard therapy that they are receiving.
  Interventions: Device: ThermoNeuroModulation TNM Device
- Sham CVS Group (Sham Comparator): In this arm participants will receive 5 sessions of twice daily sessions of 15 minutes of sham stimulation with the ThermoNeuroModulation TNM Device. The ThermoNeuroModulation TNM device will be fitted and turned on in a random paradigm that has no demonstrated efficacy. Participants will continue with the standard therapy that they are receiving.
  Interventions: Device: ThermoNeuroModulation TNM Device

INTERVENTIONS:
Device: ThermoNeuroModulation TNM Device — Study participants will undergo 10 sessions 15 minutes each of Caloric Vestibular Stimulation across 5 days with the FDA approved CVS device. This will be administered in home by study coordinators. Participants will be asked to fill out ODAS, GAD-7, and PHQ-9 on each of the five days during treatment; there is the possibility that other drug specific surveys will be used. Participants will receive two approximately 1 hour MRI scans at the beginning and at the end of the study period.
  Other Names: caloric vestibular stimulation; CVS; ThermoNeuroModulationTNM Device

SUMMARY:
The purpose of this study is to determine efficacy and effect of CVS (caloric vestibular stimulation)

DETAILED DESCRIPTION:
This study is designed as a nonrandomized, single-blind, sham-controlled trail in which willing participants will receive a 5 day course of twice daily caloric vestibular stimulation (CVS) or sham treatment. CVS involves twice daily sessions of CVS each lasting 15 minutes. The week before the intervention baseline characterization of mood and substance craving will be conducted using standard mood and substance use questionnaires. Prior to treatment beginning participants will undergo structural and functional MR imaging. Participants will also undergo a standard battery of questionnaires, including cognitive testing, mood and affect surveys, and surveys specific to SUD. During each of the 5 treatment days the participants will be asked to fill out questionnaires related to mood and craving symptoms. Participants will be blinded to sham stimulation or the standard CVS protocol. At the end of the 5 day course participants will be scanned again in MRI and asked to fill out the same battery of questions. Consistent with the existing standard of care participants will also receive two urine drug screens (UDS)

ELIGIBILITY:
Inclusion Criteria:

* Subjects will have a diagnosed SUD (including but not limited to Opiate, Alcohol, Cocaine, Nicotine, or Amphetamine Use Disorders).
* Subjects will be between the age of 17 and 50 years old
* Subjects will have been abstinent on a stable treatment regimen for at least 4 weeks
* Subjects will be able to sit still for MRI imaging
* Subjects will be able to read and complete survey questionnaires
* Subjects will reliably be abstinent from their drug of choice through the 5 day intervention as determined by the discretion of a clinician

Exclusion Criteria:

* Subjects will be excluded for comorbid neuropathology (eg history of stroke or TBI)
* Subjects will be excluded if they are at high risk for relapse as determined by a clinician
* Subjects will be excluded if they are unable to tolerate the CVS devise
* Subjects will be excluded if they have malformations of or existing trauma to the external auditory canal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
ODAS score measuring craving severity | 3 months
  Measured items 5a and 5b of the ODAS (Opiate Dosage Adequacy Scale) that deal with craving and craving severity directly. It is scored by Likert-type scores ranging from 1 to 5. The higher the score the higher the craving severity A reduction in craving and craving severity will be the primary outcome. This single dimension is important for risk of relapse, but does not by itself represent treatment adequacy as a whole.
ODAS score measuring adequacy of treatment | 3 months
  Measured by ODAS (Opiate Dosage Adequacy Scale).The ODAS clinical interview includes 10 items that evaluate six components of the construct "dose adequacy." Questions on the ODAS that measure symptom frequency are coded with Likert-type scores ranging from 1 to 5. Questions that measure symptom severity are coded on a visual analogue scale (VAS) using the same score range. The dimensional model provides a total score derived from a weighted sum of the scores of the individual items. The higher the total score, the more "adequate" the dose is considered to be. An increase in the total ODAS dimensional model score will indicate improved adequacy of treatment. This adequacy includes craving, but also represents multiple dimensions relevant to the treatment of OUD. An improvement of adequacy, irrespective of craving, is indicative of an effective treatment, and would indicate an effect of treatment on a feature of OUD other than craving.

SECONDARY OUTCOMES:
GAD-7 scores measuring anxiety | 3 months
  Measured by GAD-7 questionnaire. Scale range 0-3 with lower scores denoting better outcome measures.
PHQ-9 scores measuring Depressive Symptoms | 3 months
  Measured by PHQ-9 questionnaire. Scale range 0-3 with lower scores denoting better outcome measures.

OTHER OUTCOMES:
Resting State Functional MRI | 6 months
  Blood oxygenation-level dependent signal will be assessed for the whole brain during quiet rest
Network Connectivity | 6 months
  BOLD signal correlation of regions of interest will be conducted. Secondary network statistics including small-worldness, modularity, and others will be used to describe the network architecture.
Possible Structural Changes | 6 months
  Anatomical analysis including volumetrics will be applied to anatomical MRI scans

CONTACTS AND LOCATIONS:
Overall Officials: Margaret R Rukstalis, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Black RD, Rogers LL, Ade KK, Nicoletto HA, Adkins HD, Laskowitz DT. Non-Invasive Neuromodulation Using Time-Varying Caloric Vestibular Stimulation. IEEE J Transl Eng Health Med. 2016 Oct 7;4:2000310. doi: 10.1109/JTEHM.2016.2615899. eCollection 2016. PMID 27777829
- [Background] Gonzalez-Saiz F, Lozano Rojas O, Trujols J, Alcaraz S, Sinol N, Perez de Los Cobos J; Buprenorphine Naloxone Survey Group. Evidence of validity and reliability of the Opiate Dosage Adequacy Scale (ODAS) in a sample of heroin addicted patients in buprenorphine/naloxone maintenance treatment. Drug Alcohol Depend. 2018 Feb 1;183:127-133. doi: 10.1016/j.drugalcdep.2017.10.035. Epub 2017 Dec 11. PMID 29247974
- [Background] Gurvich C, Maller JJ, Lithgow B, Haghgooie S, Kulkarni J. Vestibular insights into cognition and psychiatry. Brain Res. 2013 Nov 6;1537:244-59. doi: 10.1016/j.brainres.2013.08.058. Epub 2013 Sep 6. PMID 24012768
- [Background] Trojak B, Sauvaget A, Fecteau S, Lalanne L, Chauvet-Gelinier JC, Koch S, Bulteau S, Zullino D, Achab S. Outcome of Non-Invasive Brain Stimulation in Substance Use Disorders: A Review of Randomized Sham-Controlled Clinical Trials. J Neuropsychiatry Clin Neurosci. 2017 Spring;29(2):105-118. doi: 10.1176/appi.neuropsych.16080147. Epub 2017 Mar 15. PMID 28294707